CLINICAL TRIAL: NCT06538714
Title: Impact of Different Interval Training Protocols on Physical, Cardio-metabolic, Lipidomic, Hematological and Psychological Parameters in Young Overweight/Obese Girls
Brief Title: Interval Training and Cardio-metabolic Health in Overweight/Obese Girls
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association Tunisienne d'Etude & de Recherche sur l'Athérosclérose (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CERB 16/2024
Record Dates: First submitted 2024-06-14; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Exercise Overtraining; Enjoyment; Cardiometabolic Syndrome; Obesity
Keywords: interval training; obesity; overweight; childhood; cardiometabolic risk; enjoyement; lipidomics; body composition; physical fitness
MeSH Terms: conditions — Overtraining Syndrome; Metabolic Syndrome; Obesity; Overweight | interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MIIT (Experimental): 12-week supervised exercise program consisting of moderate -intensity interval training (MIIT)
  Interventions: Other: MIIT
- MIIT+ HIIT (Active Comparator): 12-week supervised exercise program consisting of moderate-intensity interval training (MIIT) (6-week) and high-intensity interval training (HIIT) (6-week).
  Interventions: Other: MIIT + HIIT
- Control group No training (Placebo Comparator)
  Interventions: Other: Control group

INTERVENTIONS:
Other: MIIT — 12-week supervised exercise program consisting of moderate-intensity interval training (MIIT)
  MIIT: 3 series of 4-8 repetitions of 30-s of work at 70-75% of MAS and 30-s of active recovery at 50% of MAS.
  3 exercise sessions per week.
  Additionally, participants receive no individualized nutritional counseling.
  Arms: MIIT
Other: MIIT + HIIT — 12-week supervised exercise program consisting of moderate-intensity interval training (MIIT) (6-week) and high-intensity interval training (HIIT) (6-week).
  MIIT: 3 series of 4-8 repetitions of 30-s of work at 70-75% of MAS and 30-s of active recovery at 50% of MAS.
  HIIT: 3 series of 5 repetitions of 30-s of work at 100% of MAS and 30-s of active recovery at 50% of MAS for weeks 7-9, as well as two series of 10 repetitions of 30-s of work at 100% of MAS and 30-s of active recovery at 50% of MAS for weeks 10-12.
  3 exercise sessions per week. Additionally, participants receive no individualized nutritional counseling.
  Arms: MIIT+ HIIT
Other: Control group — Habitual physical activity No additional physical intervention
  Additionally, participants receive no individualized nutritional counseling.
  Arms: Control group No training

SUMMARY:
The main purpose of this study is to compare the impact of 12-week moderate-intensity interval training (MIIT) versus combined MIIT with high-intensity interval training (HIIT) on physical fitness, cardio metabolic, lipidomic, hematological and psychological characteristics in young overweight/obese girls.

ELIGIBILITY:
Inclusion Criteria:

* Female gender,
* Overweight or obese according to the BMI classification,
* Age, 12 to 15 years,
* Personal or parental/guardian written consent

Exclusion Criteria:

* Severe infectious or inﬂammatory diseases,
* Irregular menstrual cycles
* Participation in organized exercise training in the last 6 months or additional physical -
* recreational activities, except physical education classes.
* Using medications, hormone therapy or dietary supplements

Ages: 12 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-08-19 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | 12 weeks
  measures of weight in kilograms, height in meters, calculation of BMI in kg/m^2)
Changes in plasma triglycerides | 12 weeks
  will be assessed using an Alinity-Abbott autoanalyzer
Enjoyment | 6 and 12 weeks
  Enjoyment will be measured using the validated Physical Activity Enjoyment Scale. This scale was used to assess the level of enjoyment following interventions using the participants' responses to 18 items rated on a 7-point bipolar rating scale. The assessment consists of questions relateding to the enjoyment after intervention with the instruction, "Please rate how you feel about the physical activity you have been doing at the moment about the physical activity you have been doing". An overallOverall enjoyment of physical activity score was generated by summing the individual item scores. Scores ranged from 18-126, with higher scores reflecting higher levels of enjoyment.

SECONDARY OUTCOMES:
Changes in Aerobic velocity | 6 and 12 weeks
  Aerobic velocity will be measured with incremental running test "the Spartacus test". This test is validated for the evaluation of aerobic capacity for obese adolescents. A rectangle of 750 m (75 × 10 m) will be created with different marks set at regular intervals, which represent the different speeds (from 7 to 18 km/h). Each stage lasts three minutes whereby the first stage is set at 7 km/h and each following stage increasing by 1 km/h. During each stage, the participant had 15 s to reach the corresponding mark and then 15 s of rest. Participants adjusted their running speed simultaneously to cones and audio beep. The test ended when the subject was no longer able to maintain the pace for two consecutive occasions or when he decided to stop due to exhaustion.
Changes in lipidomic profile | 12 weeks
  Lipidomic profile will be assessed by measuring selected plasma polyunsaturated fatty acids (PUFAs), oxylipins and endocabnnabinnoids by LC-MS/MS method
Changes in hematological parameters | 12 weeks
  Hematological parameters included red blood cell count, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, leukocyte count , neutrophil count , lymphocyte count, monocyte count , eosinophil count and platelet count will be measured using an automated cell counter (Sysmex XN450; Norderstedt, Germany).
Change in Heart rate | 12 weeks
  Heart rate will be recorded using a heart rate monitor (S810, Polar, Kempele, Finland) during the incremental running test "the Spartacus test".
Change in sprint performance | 12 weeks
  Sprinting performance will be evaluated by 10-m, 20-m, 30 --m and 60-m sprints, using a series of paired photocells with an accuracy of 0.01 s (Brower Timing System, Salt Lake City, UT).

CONTACTS AND LOCATIONS:
Locations (2):
- Tunisia (2):
  - ATERA : Association Tunisienne d'Etude & de Recherche sur l'Athérosclérose, Tunis
  - Rabta Hospital, Tunis

IPD SHARING:
Plan to Share IPD: Undecided